CLINICAL TRIAL: NCT05024370
Title: Multiparas Attitude to Outpatient Care After Cesarean Section - A Qualitative Study
Brief Title: Multiparas Attitude to Outpatient Cesarean Section
Status: Completed | Type: Observational
Sponsor: Herning Hospital (Other)
Responsible Party: Principal Investigator, Iben Lorentzen, Midwife, Herning Hospital
Other Study IDs: outpatientcesareanQual
Record Dates: First submitted 2014-02-24; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Postpartum Complication
Keywords: qualitative; planned cesarean section; outpatient care; Multiparas attitude

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multiparas, planned cesarean section: Multiparas having a planned cesarean section at the departement of Obstetrics and Gynecology in Herning Hospital. Uncomplicated pregnancy that makes early discharge possible.

SUMMARY:
The main purpose of this study is to explore multiparas attitude to outpatient care after a planned cesarean section.

DETAILED DESCRIPTION:
This qualitative study should provide information about:

* Multiparas reflections in relation to prefer inpatient care after a planned cesarean section
* Womens anticipation of having inpatient care after cesarean section
* The womens experiences in relation to a planned cesarean birth and the first postnatal weeks

ELIGIBILITY:
Inclusion Criteria:

* Planned elective cesarean section of multiparous women
* Singleton pregnancy
* Age of at least 18
* Gestational age between 37 and 42 weeks

Exclusion Criteria:

* Lack of consent
* Women with no or little understanding of Danish and ability to speak Danish.
* Allergies to medicine included in the pain management regimes
* Expected maternal or neonatal complications after delivery
* Birth weight of less than 2500 grams

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mulitparas having a planned cesarean section at the department of Obstetrics and Gynecology at Herning Hospital
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
womens attitude an reflections about based on interviews | october 2013- june 2014

OTHER OUTCOMES:
womens attitude and reflections | october 2013- june 2014
  this study is based on 20 interviews with 10 multiparas having a planned cesarean section. The first interview is performed about one month before term and the second interview about two weeks after the cesarean section.

CONTACTS AND LOCATIONS:
Overall Officials: Iben P Lorentzen, Midwife, Principal Investigator — Department of Obstetrics and Gynecology, Herning Hospital
Locations (1):
- Aarhus University, Aarhus, Denmark